CLINICAL TRIAL: NCT04549402
Title: Efficacy of a Physiotherapy Intervention Through Movement Visualization in Pain Management in Patients With Hemophilic Arthropathy. Randomized Multicenter Clinical Study.
Brief Title: Movement Visualization in Pain Management in Patients With Hemophilic Arthropathy.
Acronym: HeMirror
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HeMirror
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Haemophilia
Keywords: Hemophilic arthropathy; Educative intervention; Pain; Quality of life; Anxiety; Stress
MeSH Terms: conditions — Hemophilia A; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror Therapy group (Experimental): The intervention will consist of the visualization of movement through the Mirror Therapy VR® application, broadcast on a mobile device and visualized with virtual reality glasses. The knee extension and ankle dorsiflexion movements (quadriceps and sural triceps), together with the elbow flexion (elbow flexors) will be the movements to be performed, based on their functional need (walking and feeding, respectively).
  Interventions: Other: Mirror Therapy group
- Video group (Active Comparator): The intervention will consist of the visualization of movement through the reproduction of an immersive 360º video broadcast on a mobile device and viewed with virtual reality glasses. Knee extension and ankle dorsiflexion movements (quadriceps and sural triceps), together with elbow flexion (elbow flexors) will be the movements to be performed, based on their functional need (ambulation and feeding, respectively).
  Interventions: Other: Video group
- Control group (No Intervention): Patients included in the control group will not receive any physiotherapy intervention. They will continue with their routine prior to the beginning of the study.

INTERVENTIONS:
Other: Mirror Therapy group — The intervention protocol will be carried out under the same environmental conditions and, as far as possible, on time. The intervention will last 4 weeks, with a periodicity of 7 weekly sessions. In total there will be 28 sessions lasting between 15 and 45 minutes depending on the number of joints affected.
  Arms: Mirror Therapy group
Other: Video group — The intervention protocol will be carried out under the same environmental conditions and, as far as possible, on time. The intervention will last 4 weeks, with a periodicity of 7 weekly sessions. In total there will be 28 sessions lasting between 15 and 45 minutes depending on the number of joints affected.
  Arms: Video group

SUMMARY:
Background. The recurrence of hemarthrosis in patients with hemophilia favors the development of a progressive, degenerative intra-articular lesion (hemophilic arthropathy). Pain is one of the main clinical manifestations of this arthropathy.

Objective. Assess the safety and efficacy of a pain intervention by visualizing movement using an augmented reality mobile application and immersive 360º video, regarding the frequency of bleeding and the improvement in pain perception and quality of life, joint condition , strength and functionality in patients with hemophilic arthropathy.

Study design. Randomized, multicenter, single-blind clinical study. Method. 70 patients with hemophilia A and B will be recruited in this study. The patients will be recruited in 5 regions of Spain. The 8 dependent variables will be: frequency of bleeding (self-registration), pain (measured with the visual analog scale and pressure algometer, Tampa Scale of Kinesiophobia and Pain Catastrophizing Scale), quality of life (SF-12 scale), anxiety (questionnaire of Anxiety Status-Trait-STAI), joint status (Hemophilia Joint Health Score scale), muscle strength (dynamometer) and functionality (6-Minutes Walking test, Quick Disabilities of the arm, shoulder and hand). Three evaluations will be carried out: pre-treatment, post-treatment and after a follow-up period of 6 months.

Expected results. To observe the efficacy of the visualization of movement in the characteristics of pain, and its implication in the functionality, joint state, muscular strength and the perception of quality of life in patients with hemophilic arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* Patients with a medical diagnosis of hemophilic arthropathy and pain
* People over 18 years of age
* Patients on prophylactic or on-demand treatment regimen with FVIII / FIX concentrates

Exclusion Criteria:

* Patients with neurological or cognitive disorders that impede understanding of the questionnaires
* Pain free patients
* Amputees, epileptics or patients with severe vision problems
* Patients who are receiving Physiotherapy treatment at the time of the study
* Patients who have not signed the informed consent document

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline hemarthrosis after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  A self-registration will be used to evaluate the frequency of bleeding, and thus the safety of the technique. This self-registration will be given to each patient at the beginning of the study and they must fill in the number of hemarthrosis and their main characteristics: date, origin (traumatic or spontaneous) and location (knee, ankle or elbow). The self-registration will be delivered to the evaluator in each of the study evaluations (post-treatment and follow-up).

SECONDARY OUTCOMES:
Change from baseline joint pain after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  The visual analog scale will be used to assess the perception of joint pain, being valued with a range of 0 to 10 points (from no pain to the maximum pain suffered or imaginable) in the joints evaluated
Change from baseline pressure pain threshold after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  With a pressure algometer (model Wagner FPN100) we will measure the pressure pain threshold, at the joint level and at a distance (in another part of the body). This device measures in Newton / cm2 the pressure at which the subject perceives pain under pressure. A pressure will be made on the chosen point, which we will increase at an approximate speed of 50kPa / s until the patient warns us that the sensation begins to be painful. Hemophilic arthropathy will be assessed in the elbow (on the lateral epicondyle, in the C5-C6 joint and in the tibialis anterior muscle), knee (inner edge of the patella, and tibialis anterior and extensor carpi longus muscles) and ankle (lateral malleolus, L5 spinous process, and extensor carpi longus muscle).
Change from baseline muscle strength after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  With a pressure dynamometer (microFET®2 Digital Handheld model) we will measure the strength of the biceps brachii, quadriceps and triceps surae. This device measures in Newton the force that the patient exerts in the requested muscular action. The higher the value, the greater the muscle strength. We will carry out the measurements bilaterally. The patient will be asked 4 maximum isometric contractions of 5 seconds, with a rest of 30 seconds between them, against the dynamometer located in the hand of the evaluator
Change from baseline electrical activity of the muscles after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Using surface electromyography (model SHIMMMER2, Shimmer, Ireland), we will evaluate the electrical activity of the musculature and its level of activation. The placement of the electrodes will be marked on the standing subjects, and they will be placed following the European recommendations for the use of the SEMG. A bipolar SEMG system will be used with circular electrodes 10 mm in diameter, 20 mm apart, placed longitudinally, in the direction of the fibers of the studied muscle, and with a remote reference electrode.
Change from baseline perception of quality of life after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  Using the generic Short Form 12 (SF-12v2) scale, the perception of quality of life of the patients included in the study will be evaluated. This scale consists of 12 items and a range from 0 to 100 points (where a higher score indicates a better perception of quality of life).
Change from baseline perception of anxiety after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  With the State-Trait Anxiety Inventory (STAI) scale, the perception of anxiety of the patients included in the study will be measured. The state and the anxiety trait of each subject are evaluated with a score of 0 to 30 points for each scale, where a higher score indicates a higher anxiety index in the trait or state.
Change from baseline kinesiophobia after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  With the Tampa Scale of kinesiophobia (TSK-11SV) questionnaire, the fear of movement of the patients included in the study will be evaluated. It consists of 11 items. Its values have a range of 1 to 4 points, where the higher the score, the greater the fear of movement.
Change from baseline catastrophizing after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  With the Pain catastrophizing scale questionnaire, the catastrophizing of patients with congenital coagulopathies will be measured. The scale, made up of 13 items, is assessed with a range of 0 to 4 points (lower score indicates less catastrophism).
Change from baseline joint status after treatment and at 2 months | Screening visit, within the first seven days after treatment and after two months follow-up visit
  With the Hemophilia Joint Health Score scale, specific for its use in patients with hemophilia, the joint status of patients with hemophilic arthropathy will be evaluated. It evaluates 8 items: inflammation and duration of this, pain, muscle atrophy and strength, crackles, and loss of flexion and extension. It has a score of 0 (no joint damage) to 20 points (maximum joint damage) per joint (elbows, knees and ankles). A gait rating is added to the 120 points (range 0-4 points), the maximum rating on this scale being 124 points.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- European University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No